CLINICAL TRIAL: NCT03188263
Title: Morning Light Treatment at Home to Improve Glucose Metabolism in People at Increased Risk for Type 2 Diabetes
Brief Title: Morning Light Treatment to Improve Glucose Metabolism
Acronym: ML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Rush University (Other)
Responsible Party: Principal Investigator, Kristen Knutson, Associate Professor, Center for Circadian and Sleep Medicine, Department of Neurology, Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00204710
Record Dates: First submitted 2017-06-01; First posted 2017-06-15 (Actual); Results first posted 2020-12-29 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: PreDiabetes; Circadian Dysregulation
Keywords: diabetes; sleep; circadian rhythm; light treatment
MeSH Terms: conditions — Prediabetic State; Chronobiology Disorders; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: half will receive active light treatment device, the other half will receive a placebo device
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright Light (Experimental): Irradiance is 230 μW/m2 and lux is 500 lux.
  Interventions: Other: Bright Light
- Dim Light (Placebo Comparator): irradiance is reduced from 230 μW/m2 to 3 μW/m2, and lux reduced from 500 lux to 7 lux
  Interventions: Other: Dim Light

INTERVENTIONS:
Other: Bright Light — 1 hour daily morning light treatment provided through a head-worn device for 4 weeks with the following settings: irradiance is 230 μW/m2 and lux is 500 lux.
  Arms: Bright Light
Other: Dim Light — 1 hour daily morning light treatment provided through a head-worn device for 4 weeks with the following settings: irradiance in this dimmed is reduced from 230 μW/m2 to 3 μW/m2, and lux reduced from 500 lux to 7 lux
  Arms: Dim Light

SUMMARY:
The primary purpose of this pilot study is to test a novel head worn light device (Re-Timer®) as an intervention to improve glucose metabolism in people with prediabetes. The hypothesis is that morning light treatment will improve glucose metabolism. This is a pilot study and the data from this project will be used to develop a larger clinical trial.

DETAILED DESCRIPTION:
This is a pilot study to determine whether light treatment can improve glucose metabolism in people with prediabetes. Individuals will be asked to complete a baseline session with one-week of at-home sleep monitoring followed by a 24-hour stay in the clinical research unit. During this stay, we will sample saliva in the evening to measure melatonin to estimate the timing of the internal biological clock ("circadian phase") and then we will perform a 3-hour oral glucose tolerance test in the morning to estimate markers of glucose metabolism, including insulin sensitivity. The participants will then be given a light device and instructed on its use. They will use the device for four weeks and visit our laboratory every week for a check-in. At the end of the four weeks, they will repeat the 24-hour stay in the clinical research unit.

ELIGIBILITY:
Inclusion Criteria: 34 subjects (50% female, age 40-65 y)

Subjects will be:

* Prediabetic (HbA1c 5.7% to <6.5%)
* overweight or obese (BMI>25 kg/m2)
* be free of moderate to severe obstructive sleep apnea (apnea-hypopnea index<30).

The laboratory sessions will occur during women's follicular phase or women will be postmenopausal (≥6 months since last menses).

Subjects will be scheduled to participate ≥ 1 month from travel outside the central time zone, and during a time with minimal special events.

Exclusion Criteria:

* Women who are pregnant, planning on becoming pregnant, or are breastfeeding.
* Women on oral contraceptives or hormone replacement therapy will be excluded (alters OGTT and melatonin).
* Men and women who have a child at home that does not sleep through the night will be excluded.
* Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, and prisoners are also excluded.
* History of any form of diabetes, including use of diabetes medications
* Age outside 35-70 years (we will not enroll anyone older than 70 years because of a reduced response to light).
* Smokers
* Shift workers
* Failed urine drug test (drugs of abuse, nicotine)
* Eye disease/photosensitizing medications
* Sleep medications, diagnosed sleep disorders (history of treatment may affect glucose metabolism),
* Daily beta-blocker, NSAID or melatonin use (confounds DLMO)
* History of psychiatric disorders (confounds effect of light treatment, per relevant items from Mood Disorder, Psychotic Screening and Substance Use Disorders Modules of the Structured Clinical Interview for DSM-IV Axis I Disorders - Non-Patient Edition (SCID-IV/NP) to screen for schizophrenia, bipolar depression, substance abuse, suicidal ideation, obsessive compulsive disorder, PTSD), depressive symptoms using the Center for Epidemiologic Studies - Depression (CES-D) scale
* Irregular menses
* History of cardiovascular disease (excluding hypertension), endocrine, kidney, gastrointestinal or liver disorder, seizures, and cancer.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Knutson, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bright Light | Dim Light
Started | 10 | 0
Completed | 6 | 0
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were no participants enrolled into the dim light condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bright Light | Dim Light | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 9 |  | 9
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (8.0) |  | 52.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  | 6
  Male | 4 |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 8 |  | 8
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 7 |  | 7
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 |  | 10
Hemoglobin A1c (%), Continuous [Mean (Standard Deviation); unit: % of hemoglobin bound to glucose] | 6.0 (0.2) |  | 6.0 (0.2)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 34.5 (7.1) |  | 34.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glucose Levels (Area-under-the-curve) Measured by Performance on Oral Glucose Tolerance Test (OGTT)
Description: The OGTT is a 3-hour procedure measuring blood glucose levels after the patient has consumed a 75-gram dextrose solution at -15 min, 0 min, 30 min, 60 min, 90 min, 120 min, and 180 min intervals. Total area-under-the-curve of glucose levels is calculated.
Time Frame: Change from baseline to after 4 weeks of light treatment
Population: There were no participants enrolled into the dim light condition.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Bright Light | Dim Light
Number analyzed (Participants) | 6 | 0
mg*h/dL | -11.3 (11.0) |
Statistical Analysis 1: Comparison: Bright Light; The primary planned analyses was to examine effect in bright light group. A significance level of .05 was selected a priori; Test type: Other — The primary planned analysis was in bright light group only and compared pre-post measurements; p = .046, Sign test — A threshold of .05 was selected a priori; A Wilcoxon matched-pairs signed-ranks test was estimated to determine if pre-post measures of glucose levels differed significantly

2. Secondary Outcome: Changes in Circadian Phase Measured by Dim Light Melatonin Onset (DLMO)
Description: The DLMO is measured via saliva samples collected during laboratory sessions. A sample is collected every half hour until bedtime starting 6.5 hours before habitual bedtime, and conducted in dim light setting to identify the point when melatonin starts being released.
Time Frame: Change from baseline to after 4 weeks of light treatment.
Population: There were no participants enrolled into the dim light condition. In addition, one participant in the bright light condition was missing a valid DLMO measurement.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bright Light | Dim Light
Number analyzed (Participants) | 5 | 0
hours | -0.6 (1.9) |
Statistical Analysis 1: Comparison: Bright Light; [analysis description as in outcome 1, analysis 1]; Test type: Other — The primary planned analysis was in bright light group only and compared pre-post measurements; p = .35, Sign test — A threshold of .05 was selected a priori; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: There were no participants enrolled in the dim light group and therefore there was no one at risk.
Arm/Group | Bright Light | Dim Light
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/0

LIMITATIONS AND CAVEATS:
Our planned enrollment goal was 14 participants in each group and therefore we were underpowered in the bright light group to detect changes in all outcome measures. Further, we were not able to perform secondary analyses, which included between group comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT03188263/Prot_SAP_ICF_000.pdf